CLINICAL TRIAL: NCT00334074
Title: Phase II Trial of Clofarabine and Cytarabine in Relapsed Standard-Risk AML and Untreated High-Risk MDS in Adult Patients, and Untreated AML in Selected Elderly Patients at High Risk of Anthracycline Toxicity
Brief Title: Clofarabine and Ara-C for the Treatment of Relapsed AML and Untreated MDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 004-145; 004-145 (Other: Baylor Internal Review Board)
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Results first posted 2013-07-17 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndromes; Chronic Myelogenous Leukemia
Keywords: AML; MDS; CML; Relapsed; Refractory; Chemo treatment; Clofarabine; Cytarabine; standard or poor cytogenetic risk AML; untreated high-risk (>10% blasts) MDS; CML in accelerated phase or blast crisis; Elderly AML patients with risk of anthracycline toxicity
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Recurrence; Blast Crisis | interventions — Clofarabine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clofarabine and Cytarabine (Experimental): Five consecutive days of clofarabine 40 mg/m^2 IVI over 1 hour followed 4 hours later by cytarabine 1000 mg/m^2 IVI over 2 hours
  Interventions: Drug: Clofarabine and Cytarabine

INTERVENTIONS:
Drug: Clofarabine and Cytarabine — Phase II Trial of Clofarabine and Cytarabine in Relapsed Standard-Risk AML and Untreated High-Risk MDS in Adult Patients, and Untreated AML in selected Elderly Patients at high risk of anthracycline toxicity
  Other Names: Clofarabine: CAFdA; Cl-F-ara-A; Cytarabine: Ara-C

SUMMARY:
The purpose of this trial is to to determine the safety and effectiveness of therapeutic combination - Clofarabine and Cytarabine for the treatment of AML and MDS.

DETAILED DESCRIPTION:
Previous studies of Clofarabine and Cytarabine combination treatment in adult AML and MDS patients showed promising results.

This study is done to confirm the findings from previous studies. Primary objective is to determine the overall response rate (complete response [CR] plus partial response [PR]); secondary objective of this study is to characterize and quantify the toxicity profile associated with clofarabine plus cytarabine treatment.

A maximum of 35 patients will be treated on this study. They will receive 5 consecutive days of clofarabine intra venous infusion (IVI) followed 4 hours later by cytarabine IVI.Patients will receive up to a maximum of 4 cycles of study treatment. Next cycle will start approximately 4 weeks after Day 1 of previous cycle.No other investigational or commercial agents including chemotherapy, radiotherapy, or immunotherapy may be administered to patients enrolled in this study with the intention of treating the underlying malignancy

Patients will remain on study, and be monitored until 4 months have elapsed from the beginning date of their last cycle of treatment.

ELIGIBILITY:
Adult patients who are at least 18 years old with histologically confirmed disease as follows:

* Standard or poor cytogenetic risk acute myelogenous leukemia (AML) according to the Southwestern Oncology Group (SWOG) criteria in first relapse or primary refractory status
* Untreated high-risk myelodysplastic syndrome (MDS) defined as >10% blasts
* Chronic myelogenous leukemia (CML) in accelerated phase or blast crisis failing imatinib therapy.
* Selected elderly patients with untreated AML who are at high risk of anthracycline toxicity.

Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or
* Laboratory values obtained less than or equal to 7 days prior to receiving study treatment:

  * Total bilirubin < 2.0 mg/dL unless elevated due to hemolysis
  * Aspartate transaminase (AST)/alanine transaminase (ALT) less than or equal to 5 × upper limit of normal (ULN)
  * Serum creatinine < 2.0 mg/dL
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent.
* Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment.
* Male and female patients must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment.

Exclusion Criteria:

* Patients with FAB M3 unless relapsed after treatment with ATRA and arsenic trioxide.
* Patients eligible to receive curative allogeneic transplant as determined by performance status, organ function, availability of a matched donor, etc.
* Current concomitant chemotherapy, radiation therapy, or immunotherapy.
* Use of investigational agents within 30 days or any anticancer therapy within 3 weeks before study entry. The patient must have recovered from all acute toxicities from any previous therapy.
* Active heart disease including myocardial infarction within the preceding 3 months.
* History of severe coronary artery disease, arrhythmias other than atrial flutter or fibrillation requiring medication, or uncontrolled congestive heart failure
* Dyspnea at rest or with minimal exertion.
* Patients with an active, uncontrolled systemic infection considered to be opportunistic, life-threatening, or clinically significant at the time of treatment or with a known or suspected fungal infection (ie, patients on parenteral antifungal therapy).
* Pregnant or lactating patients.
* Prior enrollment in this trial.
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-08; Primary Completion 2007-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Agura, MD, Principal Investigator — Baylor University Medical Center - Director Blood and Marrow Transplantation Services
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited after the initial IRB approval in september 2004 at Baylor University Medical Center. Enrollment was closed in october 2006. The study was completed Including follow up in February 2007.
Groups:
- Clofarabine and Cytarabine: 5 consecutive days of Clofarabine 40 mg/m^2 intravenous infusion over 1 hour followed 4 hours later by cytarabine 1000mg/m^2 intravenous infusion over 2 hours.Next cycle will start approximately 4 weeks after Day 1 of previous cycle. Patients will receive a maximum of 4 cycles of study treatment.
Period: Overall Study
Arm/Group | Clofarabine and Cytarabine
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Clofarabine and Cytarabine: Clofarabine 40 mg/m2 IV infusion over 1 hour for 5 days; Cytarabine 1000 mg/m2 IV infusion 4 hours post clofarabine IVI.
Arm/Group | Clofarabine and Cytarabine
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 64 (21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Complete Response [CR] Plus Partial Response [PR]) of Clofarabine Plus Cytarabine in Patients With Relapsed/Refractory AML, Untreated MDS, CML in Blast Phase, or in Selected Untreated Patients With High Risk of Anthracycline Toxicity
Description: Based on International working group for diagnosis, standardization of response criteria, and treatment outcomes for reporting standards for therapeutic trials in Acute myeloid Leukemia:
  Complete Response (CR) was defined as normalization of marrow blasts (< 5%), recovery of normal heamtopoiesis (absolute neutrophil count >1 X 10^9/l, platelet count ≥100 X10^9/l, and absence of peripheral blood blasts, independent of transfusions and growth factor support.
  Partial response was defined as blood count recovery as for complete response with the exception of leukemic marrow blasts in the range of 6%-25% or a ≥50% decrease in bone marrow blasts.
  Treatment failure was defined as a <25% change in marrow blasts within 30 days of starting therapy
Time Frame: Proportion of confirmed responses was estimated by the number of patients who achieved a CR or PR, defined as two consecutive evaluations at least 4 weeks apart, divided by the number of eligible participants in the study.
Population: Intent to Treat analysis; per eligible participants enrolled in the study.
Measure: Number; unit: participants
Groups:
- Clofarabine Plus Cytarabine: Clofarabine 40 mg/m2 IV infusion over 1 hour for 5 days; Four hours post clofarabine infusion,Give cytarabine 1000 mg/m2 IV infusion over 2 hours.Patients will receive a maximum upto 4 cycles of study treatment.Next cycle will start approximately 4 weeks after Day 1 of previous cycle.
Arm/Group | Clofarabine Plus Cytarabine
Number analyzed (Participants) | 30
participants
  Overall Response Rate | 16
  Complete Response | 14
  Partial Response | 2
  Not Responding | 8
  Not evaluable | 6

2. Secondary Outcome: Number of Participants Who Had an Adverse Event While on Treatment With Clofarabine Plus Cytarabine
Description: Patients will be monitored clinically and diagnostically using measures including blood test, bone marrow aspiration and MUGA. Toxicity assessment every week using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 will be performed.
Time Frame: Up to five months (includes follow up period of 30 days) from the day patient received their first dose of study drug
Population: Intention To Treat
Measure: Number; unit: participants; with adverse events
Arm/Group | Clofarabine and Cytarabine
Number analyzed (Participants) | 30
participants; with adverse events | 30

ADVERSE EVENTS:
Time Frame: 1 year 6 months. Initial IRB approval in 9/2004. Enrollment start date - 8/2005. Study completion including follow up - Feb 2007.
Groups:
- Clofarabine and Cytarabine: Clofarabine 40 mg/m2 intravenous infusion over 1 hour for 5 days; Cytarabine 1000 mg/m2 intravenous infusion 4 hours post clofarabine IVI.
Arm/Group | Clofarabine and Cytarabine
Serious Adverse Events (participants affected / at risk) | 30/30
Other Adverse Events (participants affected / at risk) | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine and Cytarabine (N=30)
Atrial Fibrillation (Cardiac disorders) | 3 (3)
Edema/Weight Gain (Blood and lymphatic system disorders) | 3 (3)
Elevated LFT (Investigations) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 2 (2)
Fever (Infections and infestations) | 3 (3)
Fungal Pneumonia (Infections and infestations) | 2 (2)
Hand and Foot Syndrome (Skin and subcutaneous tissue disorders) | 3 (3)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 24 (24)
Platelet Allosensitization (Blood and lymphatic system disorders) | 1 (1) — 1
Sepsis (Infections and infestations) | 5 (5)
Small Bowell Obstruction (Gastrointestinal disorders) | 1 (1)
Staph Bacteremia (Infections and infestations) | 1 (1)
Staph epidermitis (Infections and infestations) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Volume Overload (Blood and lymphatic system disorders) | 1 (1)
Bilateral External Otitis (Infections and infestations) | 1 (1)
Delirium (Nervous system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Multiple System Organ Failure (Infections and infestations) | 6 (6)
Perianal Abcess (Gastrointestinal disorders) | 1 (1)
Pulmonary Infiltrate (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal Insufficiency / Failure (Renal and urinary disorders) | 3 (3)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine and Cytarabine (N=30)
Diarrhea (Gastrointestinal disorders) | 17 (17)
Fever (Infections and infestations) | 13 (13)
Nausea (Gastrointestinal disorders) | 12 (12)
Rash (Skin and subcutaneous tissue disorders) | 13 (13)
Edema/Weight Gain (Blood and lymphatic system disorders) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less